CLINICAL TRIAL: NCT00002036
Title: Phase I Safety Study of Anti-HIV Immune Serum Globulin (Human)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Purpose: Treatment
Other Study IDs: 060A; 0001-008
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Immunization, Passive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex

INTERVENTIONS:
Drug: Anti-HIV Immune Serum Globulin (Human)

SUMMARY:
To investigate the potential benefit of providing passive immunity with hyperimmune anti-HIV human serum.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Proof of HIV infection.
* Diagnosis of asymptomatic HIV infection or early AIDS related complex (ARC) with no zidovudine (AZT) or other anti-HIV therapy. OR a diagnosis of AIDS and = or > 3 months of AZT therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* HIV-induced neurological disease.
* IgA negative.

Concurrent Medication:

Excluded:

* Immunomodulating agents.
* Steroids.
* Interferons.

Patients with the following are excluded:

* Active substance abuse.
* Use of immunomodulating drugs such as steroids or interferons.
* HIV-induced neurological disease.
* IgA negative.

Required with a diagnosis of AIDS:

* = or > 3 months of zidovudine (AZT) therapy.

Active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12

CONTACTS AND LOCATIONS:
Locations (1):
- Univ of Minnesota, Minneapolis, Minnesota, United States